CLINICAL TRIAL: NCT03807102
Title: Phase I/II Trial of Tumor Vaccine in Post Radical Operation Patients With Lung Cancer
Brief Title: Trial of Tumor Vaccine Used for Adjuvant Therapy in Post Radical Operation Patients With Lung Cancer
Acronym: TVATLC01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yongchang Zhang (Other)
Collaborators: Shanghai Houchao Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, MD, pHD, Director of Thoracic Surgery Department II, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVATLC01
Record Dates: First submitted 2019-01-04; First posted 2019-01-16 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cancer Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Vaccine (Experimental): Injection of NeoAntigen Tumor Vaccine
  Interventions: Biological: Tumor Vaccine

INTERVENTIONS:
Biological: Tumor Vaccine — NeoAntigen Tumor Vaccine (5 injections for each 3 days and then 1 injection for each 3 months till recurrence or up to 2 years).

SUMMARY:
Tumor vaccines may make the body build an immune response to kill tumor cells. This research study is evaluating a new type of tumor vaccine termed as "Neoantigen Tumor Vaccine". The purpose of this phase I/II trial study is to assess the safety and effectiveness of neoantigentumor vaccine in post radical operation patients with stage IIIA lung cancer.

DETAILED DESCRIPTION:
Outline: After successful vaccine manufacturing, patients receive neoantigen tumor vaccine hypodermically (5 injections for each 3 days and then 1 injection for each 3 months till recurrence or up to 2 years). Treatment continues in the absence of disease recurrence and metastasis or unacceptable toxicity.

Patients are followed for 2 years or up to the absence of disease recurrence and metastasis.

Projected accrual: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years, Male or Female
* Histological or cytologically diagnosis of lung adenocarcinoma
* After surgical treatment (lobectomy and systematic lymph node dissection)
* Pathological stage IIIA (According to the IASLC Lung Cancer Staging (eight Edition))
* Postoperative standard treatment (platinum-based double-drug adjuvant treatment with or without chemotherapy) or no adjuvant treatment
* Have potential dynamic tumor biomarkers
* Able and willing to give witnessed, written informed consent form prior to receiving any study related procedure, agree to participate in long-term follow-up for up to 3 years

Exclusion Criteria:

* Age < 18 or< 70 years
* Lung squamous cell carcinoma, small cell lung cancer, large cell lung cancer
* Without surgical treatment
* Pathological stage I、II、IIIB、IIIC or IV (According to the IASLC Lung Cancer Staging (eight Edition))
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study vaccine
* Drug or alcohol abusers
* Pregnant or breast-feeding patients
* History of immunodeficiency disease or autoimmune disease
* Patients with chronic disease which is undergoing immune reagents or hormone therapy
* Concurrent other medical condition that would prevent the patient from undergoing protocol-based therapy
* Lack of availability of a patient for immunological and clinical follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-16 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Approximately 2 years
  The time that participants stay free of cancer after surgery following administration of tumor vaccine
Adverse Events (AEs) | 30 days from first study vaccine administration
  Number of participants experiencing clinical and laboratory adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wenxiang Wang, MD, PhD, Principal Investigator — Hunan Provincal Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No